CLINICAL TRIAL: NCT02847767
Title: Dynamic Contrast Enhanced Imaging of Patients Receiving SABR for Unresectable or Medically Inoperable Hepatocellular Carcinoma in BC
Brief Title: Dynamic Contrast Enhanced HCC SABR Liver Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Principal Investigator, Francois Benard, Scientific Director, Functional Imaging, British Columbia Cancer Agency
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H15-02341
Record Dates: First submitted 2016-07-05; First posted 2016-07-28 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Liver Perfusion; Hepatocellular Carcinoma; Dynamic Contrast-Enhanced Computed Tomography
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Perfusion Imaging (Experimental): IV contrast perfusion CT will be performed at baseline and at 1 week after completing treatment. Perfusion imaging is similar to a diagnostic CT except a smaller region is serially imaged post contrast injection with multiple data acquisitions and high temporal resolution.
  Interventions: Procedure: Perfusion Imaging

INTERVENTIONS:
Procedure: Perfusion Imaging — IV contrast perfusion CT will be performed at baseline and at 1 week after completing treatment. Perfusion imaging is similar to a diagnostic CT except a smaller region is serially imaged post contrast injection with multiple data acquisitions and high temporal resolution

SUMMARY:
The high dose per fraction (>10Gy/fraction) used in Stereotactic Ablative Body Radiotherapy (SABR) has been shown to be more effective at local tumor control than treatments employing more conventional dose fractions. The mechanisms for this are currently under debate. One possible mechanism for this increased effectiveness is that high dose/fraction causes significant vascular damage to the tumor. This study hopes to measure vascular integrity pre and post SABR treatment using kinetic models obtained from dynamic contrast enhanced CT.

DETAILED DESCRIPTION:
Purpose:

The purpose of this study is to determine if high dose per fraction SABR has an impact on the vasculature of both the tumor and of healthy liver tissue.

Hypothesis:

High dose / fraction in HCC patients with tumours < 5 cm will result in detectable changes to kinetic model parameters derived from dynamic contrast enhanced images.

Objectives:

Primary objective:

To quantify changes in tumor vascular support for patients receiving SABR.

Secondary objectives:

To investigate the correlation between PK derived model liver perfusion parameters and QoL metrics as measured by EORTC QLQ-C30 and FACT-Hep QoL assessments.

Research Methods:

Target population are patients receiving liver SABR for no more than 2 discrete liver tumors with a maximum dimension <5cm.

Perfusion CT Image Data Post Processing and Analysis. Patient motion will be corrected using deformable registration, fiducial tracking, and RPM breathing traces. Organ ROIs will be added to the perfusion image series by manually translating anatomical planning CT ROIs to the motion-corrected perfusion image series, or by algorithmically deforming planning ROIs. Portal vein and abdominal aorta ROIs will be demarcated.

Analysis will proceed via custom software we have built during related projects. Contrast enhancement time courses will be generated for key structures (i.e., abdominal aorta, portal vein, and gross liver tissues) and used to derive a variety of perfusion map images, such as liver perfusion, mean transit time, arterial fraction, and distribution volume. A distributed parameter model will be preferred for kinetic modeling. Supplementary non-parametric techniques will be used for other parameters of interest (e.g., IAUC, maximum slope).

Images acquired before and after treatment will be registered so that parameter maps can be compared on a per-patient basis. Changes in perfusion parameters will be characterized with special emphasis placed on regional structure and clustering effects. Pre and post parameter maps will be computed near individual-voxel level. Regions of interest (1) within or near tumour and (2) at a low-dose portion of liver will be defined. A distribution of parameters within each ROI will be used to generate estimates of the mean parameters and uncertainty. Estimates of mean parameters and whole distributions will be compared using standard statistical comparisons (t-test and Whitney respectively).

Quality of Life We will evaluate quality of life (QOL) in HCC patients treated with SBRT using EORTC QLQ-C30 and FACT-Hep QOL assessments at baseline, 3, 6, 9 and 12 months. Correlation between perfusion parameter changes and patient outcomes or QOL (second-order analysis) will be applied if statistically significant first-order parameter changes can be detected. Standard correlative measures such as the Pearson product-moment correlation measure will be used to assess statistical significance. As there is currently no data relating liver perfusion to toxicity or quality of life, this study will examine whether a change in liver perfusion is correlated with enhanced or reduced QOL.

ELIGIBILITY:
Inclusion Criteria:

All the following criteria must be met:

1. Age > 18 years old
2. Multi-phase CT scan and/or MRI of the liver within 8 weeks of radiation planning demonstrating:

   * Liver tumours < 5 cm
   * No more than 2 discrete liver tumours
   * Normal liver > 700 cc
3. Patients must have HCC diagnosed by either: i) pathological confirmation, or ii) intrahepatic vascular enhancement of the lesion demonstrated by at least two imaging modalities, or iii) intrahepatic vascular enhancement of the lesion demonstrated by one imaging modality if AFP > 200 in the setting of liver cirrhosis or chronic hepatitis B without cirrhosis (EASL consensus guidelines [2])
4. Liver HCC must be deemed unresectable as determined by an experienced hepatobiliary surgeon, or the patient must be medically inoperable or refuse surgery,
5. Patients must be discussed in a multidisciplinary setting, with representatives from Medical Oncology, Radiation Oncology, Surgery, Interventional Radiology, and Hepatology. Patients must be considered ineligible for standard local treatments, including surgery, liver transplantation, radiofrequency ablation, and targeted biologics. Some subjects could be potential candidates for sorafenib but normally this treatment is not considered before all local treatment options have been considered, as the response rate to sorafenib is low (2% in the SHARP study). Patients might be candidates for sorafenib after progression on the study treatment or if they do not want to participate and in both cases they will be referred to a medical oncologist. Patients may have received prior TACE and had an incomplete response. Ineffective or incomplete TACE is defined as incomplete filling by lipiodol-doxorubicin mixture used by either angiography or CT ≥1 month after TACE or by increasing alpha-fetoprotein level. Patients must have recovered from the effects of previous therapies before SBRT with a minimum 4-week period between TACE and SBRT.
6. Eastern Clinical Oncology Group performance status 0, 1, or 2 (Appendix III), or a Karnofsky performance status of ≥ 60 (Appendix IV)
7. Adequate organ function as assessed by the following blood work:

   * Hemoglobin ≥ 90 g/L
   * Absolute neutrophil count ≥ 1.0 bil/L
   * Platelets ≥ 50 bil/L
   * AST and ALT not to exceed 3x upper limit of normal
8. Child-Turcotte-Pugh assessment within 8 weeks of treatment date (Appendix II):

   * Bilirubin ≤ 3 mg/dL (< 50 µmol/L)
   * Albumin above 28 g/L
   * INR < 1.7 and/or correctable with vitamin K (unless on anticoagulation therapy)
   * No ascites or encephalopathy
   * Child-Turcotte-Pugh score must be ≤ 7
9. BCLC Stage B or C (portal venous invasion or liver hilum nodal disease only; (Appendix I)
10. Life expectancy > 6 months
11. No chemotherapy or systemic therapy concurrent with radiotherapy
12. Previous treatment(s) with radiofrequency ablation, surgery, TACE, Y90, percutaneous ethanol injection, or chemotherapy are not exclusion criteria provided that recurrence or lack of tumour response has been documented. Patients who decline, or not eligible for, these treatments will also be considered eligible.
13. Patient signs a study-specific informed consent form. If the patient's mental status precludes this, written informed consent may be given by the patient's legal representative. A translator will be provided if the patient has a language barrier.
14. Treatment plans meet acceptable dose constraints and Liver Veff is ≤ 0.55

Exclusion Criteria:

1. Patients with active hepatitis, encephalopathy, or ascites related to liver failure
2. Female patients who are pregnant (verify with blood test if patient is pre-menopausal). Pre-menopausal patients may also not become pregnant during participation in this study.
3. Prior external beam radiation to the upper abdomen
4. Patients with distant metastases or extrahepatic nodal progression (patients with portal venous thrombosis and liver hilum nodal involvement remain eligible)
5. Patients who have < 700 cc of normal liver.
6. Child-Turcotte-Pugh scores > 7
7. BCLC Stage A, C (N1 and/or M1), D
8. Prior gastric, duodenal, or variceal bleed within the past 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Changes in tumour vasculature as assessed by changes PL derived model parameters | 1 week after cancer treatment
  To quantify changes in tumor vascular support for patients receiving SABR.

SECONDARY OUTCOMES:
Association (correlation) between aggregate QOL scores and PK derived model parameters | 1 week after cancer treatment
  To investigate the correlation between PK derived model liver perfusion parameters and QOL metrics as measured by EORTC QLQ-C30 and FACT-Hep QOL assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Francois Benard, MD, Principal Investigator — British Columbia Cancer Agency
Locations (2):
- Canada (2):
  - BC Cancer Agency Fraser Valley Centre, Surrey, British Columbia
  - BC Cancer Agency Vancouver Centre, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No